CLINICAL TRIAL: NCT01939106
Title: A Single Center Study to Assess the Safety and Performance of a One Piece Drainable Pouch in Subjects With an Ileostomy
Brief Title: One Piece Drainable Pouch in Subjects With an Ileostomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CC-0512-13-A740
Record Dates: First submitted 2013-07-29; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Ileostomy
Keywords: Stoma; Ileostomy; pouch; Drainable Pouch for collection of stool

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One Piece Drainable Pouch (Other): This is a one piece drainable pouch designed for the purpose of collecting stool from subjects with an ileostomy stoma
  Interventions: Device: One Piece Drainable Pouch

INTERVENTIONS:
Device: One Piece Drainable Pouch
  Other Names: Enhanced one piece drainable pouch

SUMMARY:
To assess the safety and performance of an enhanced one piece drainable pouch in subjects with an ileostomy.

DETAILED DESCRIPTION:
This is a pre market study to assess safety and performance of a one piece drainable pouch. Twelve subjects will be recruited and will use the study pouch for 10 days. During this time data on skin and stoma condition will be collected along with questions related to ease of use comfort and overall pouch performance. The study will be conducted in the US in one single site.

ELIGIBILITY:
Inclusion Criteria

1. Of legal consenting age and able to provide written informed consent
2. Is able to read, write, and understand the primary language of the investigative site.
3. Have an ileostomy for more than 3 months
4. Currently a one or two piece drainable pouch user (all attempts will be made to include ConvaTec Active Life or Esteem Plus one piece closed pouch users)
5. Have unbroken peri-stomal skin (healthy normal skin to L1 on the SACs Instrument Scale # 1)
6. Have a stoma considered 'normal' in appearance in accordance with the stoma, color, moisture and structure rating scales
7. Be willing to wear a one piece drainable pouch with moldable wafer according to the usual wear pattern of this type of pouch
8. Be willing to participate in the trial for 10 days plus 1 visit prior to the in-residence study period.
9. Be willing to remain in residence for 3 days at a central location
10. Be willing to meet with the investigator for a total of nine scheduled visits.
11. Be willing to discontinue the use of pastes, adhesive strips and rings/seals used to seal the area between the skin barrier wafer and stoma during the use of the study device
12. Other than their ileostomy considered to have a healthy/stable health status Have good manual dexterity and be able to take care of their stoma independently Be willing and able to complete a diary card for the duration of the study. Be willing to take photographs of the stoma and pouch on pouch removal

Exclusion Criteria - The following subjects must not be included into the study:

1. Subjects with a history of sensitivity to any one of the ostomy products or the components being studied
2. Subjects with stoma duration of less than 3 months
3. Subjects who currently use a belt with their usual appliance
4. Subjects who have been entered into the study before, or who have previously taken part in a study in the last month.
5. Subjects who require convexity or other skin fillers (pastes, seals, or rings) to even undulations of the peristomal skin
6. Subjects undergoing chemotherapy or radiotherapy
7. Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety | Study duration will be 10 days
  To assess the condition of the peristomal skin and stoma and number and frequency of adverse events

SECONDARY OUTCOMES:
Performance/Efficacy | The study will be for 10 days
  To assess ease of use including ease of application and removal, comfort and security along with wear time

CONTACTS AND LOCATIONS:
Overall Officials: Ann Popavich-Durnal, RN BSN, Principal Investigator
Locations (1):
- Independent Nurse Consultant LLC, Tucson, Arizona, United States